CLINICAL TRIAL: NCT01438957
Title: Phase III Randomized Placebo-controlled Double Blind Comparative Study to Investigate the Efficacy and Safety of DA-9501 in Sedation During the Surgery With Epidural Anesthesia or Spinal Anesthesia Without Intubation Under Monitored Sedation Care
Brief Title: Clinical Study to Investigate the Efficacy and the Safety of DA-9501 in Sedation During the Surgery With Epidural Anesthesia or Spinal Anesthesia Without Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Maruishi Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEX-303
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Sedation
Keywords: Dexmedetomidine; Sedation; Non-intubation; epidural anesthesia; spinal anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (5):
- Placebo (Placebo Comparator): Dexmedetomidine 0 mcg/kg/hr 10 min Initial dose + Dexmedetomidine 0 mcg/kg/hr Maintenance dose
  Interventions: Drug: Placebo
- Dexmedetomidine 0.067 mcg/kg (Experimental): Dexmedetomidine 0.4 mcg/kg/hr 10 min Initial dose + Dexmedetomidine 0.2 - 0.7 mcg/kg/hr Maintenance dose
  Interventions: Drug: Dexmedetomidine hydrochloride
- Dexmedetomidine 0.25 mcg/kg (Experimental): Dexmedetomidine 1.5 mcg/kg/hr 10 min Initial dose + Dexmedetomidine 0.2 - 0.7 mcg/kg/hr Maintenance dose
  Interventions: Drug: Dexmedetomidine hydrochloride
- Dexmedetomidine 0.5 mcg/kg (Experimental): Dexmedetomidine 3 mcg/kg/hr 10 min Initial dose + Dexmedetomidine 0.2 - 0.7 mcg/kg/hr Maintenance dose
  Interventions: Drug: Dexmedetomidine hydrochloride
- Dexmedetomidine 1.0 mcg/kg (Experimental): Dexmedetomidine 6 mcg/kg/hr 10 min Initial dose + Dexmedetomidine 0.2 - 0.7 mcg/kg/hr Maintenance dose
  Interventions: Drug: Dexmedetomidine hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine hydrochloride — Dexmedetomidine 0.2 to 0.7 mcg/kg/hr
  Arms: Dexmedetomidine 0.067 mcg/kg; Dexmedetomidine 0.25 mcg/kg; Dexmedetomidine 0.5 mcg/kg; Dexmedetomidine 1.0 mcg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy and safety of DA-9501 (Dexmedetomidine) in patients who require sedation during the surgery that requires epidural or spinal anesthesia without intubation under monitored sedation care.

DETAILED DESCRIPTION:
Phase III, randomized, placebo controlled, double blind, parallel comparative study (Therapeutic confirmatory trial), to evaluate the efficacy and the safety of Dexmedetomidine in non-intubated patients who require sedation during surgery with spinal or epidural anesthesia under monitored sedation care

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed and dated the Informed Consent after the study had been fully explained.
2. Patient is male or female, at least 20 years of age when the Informed Consent is obtained.
3. American Society for Anesthesiologists (ASA) I to III Class.
4. Patient who requires sedation during the elective surgery which requires ≥30mins (expected time) without intubation under monitored sedation care.
5. Patient undergoing a surgery requiring epidural or spinal anesthesia

Exclusion Criteria:

1. Patient who underwent general anesthesia within 7 days, or who received other study drugs within 30 days from the date of consent.
2. Patient with <92% SpO2, at the physical examination prior to the study drug administration, or ventilatory failure which requires intubation or Laryngeal Mask.
3. Patient with central nervous system pathology which may lead to increased intracranial pressure, uncontrolled seizures, psychiatric disorder which may be confused with the response to sedation treatment.
4. Patient who require general anesthesia.
5. Patient who receives treatment by alpha-2 agonists or alpha-2 antagonists within seven days of scheduled surgery or procedure.
6. Patient in whom opioids, DA-9501 or other alpha-2 agonists, or drugs which may be used in the study are contraindicated.
7. Patient diagnosed with unstable angina or acute myocardiac infarction within 6 weeks from the date of consent.
8. Patient whose heart rate is <60 bpm, systolic blood pressure is <90 mmHg by the physical examination prior to the study drug administration.
9. Patient has third degree heart block, unless the patient has a pacemaker or transverse pacing wires are in place.
10. Patient who has experienced an increase in alanine transaminase (ALT) and / or aspartate aminotransferase (AST) more than double the upper normal limit within 2 months of the date of consent, or who has a history of liver insufficiency.
11. Pregnant or lactating woman.
12. In the Investigator's or subinvestigator's opinion, the patient has any symptom or condition which might increase risk to the patient by conducting the study or preclude obtaining satisfactory study data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-06-03 (Actual); Primary Completion 2011-11-18 (Actual); Study Completion 2011-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Japan (12):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kochi Medical School Hospital, Nangoku, Kochi
  - Shinshul University Hospital, Matsumoto, Nagano
  - Shimane University Hospital, Izumo, Shimane
  - Tottori University Hospital, Yonago, Tottori
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - University of Miyazaki Hospital, Miyazaki
  - Okayama University Hospital, Okayama
  - Kitano Hospital, The Tazuke Kofukai Medical Research Institute, Osaka
  - Nippon Medical University Hospital, Tokyo

REFERENCES:
- [Derived] Inagaki Y, Yamakage M, Sakamoto A, Okayama A, Oya N, Hiraoka T, Morita K. The Efficacy and Safety of Dexmedetomidine for Sedation During Surgery Under Epidural or Spinal Anesthesia: A Randomized, Double-Blind, Placebo-Controlled Study. Yonago Acta Med. 2022 Jan 4;65(1):14-25. doi: 10.33160/yam.2022.02.002. eCollection 2022 Feb. PMID 35221757

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 0 mcg/kg/hr 10min Initial dose + 0 mcg/kg/hr Maintenance dose
- Dexmedetomidine 0.067 mcg/kg: 0.4 mcg/kg/hr 10min Initial dose + 0.2-0.7 mcg/kg/hr Maintenance dose
- Dexmedetomidine 0.25 mcg/kg: 1.5 mcg/kg/hr 10min Initial dose + 0.2-0.7 mcg/kg/hr Maintenance dose
- Dexmedetomidine 0.5 mcg/kg: 3 mcg/kg/hr 10min Initial dose + 0.2-0.7 mcg/kg/hr Maintenance dose
- Dexmedetomidine 1.0 mcg/kg: 6 mcg/kg/hr 10min Initial dose + 0.2-0.7 mcg/kg/hr Maintenance dose
Period: Overall Study
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Started | 22 | 23 | 24 | 25 | 25
Completed | 21 | 22 | 24 | 24 | 25
Not Completed | 1 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg | Total
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25 | 119
Age, Continuous [Mean (Full Range); unit: years] | 69.0 [51 to 86] | 60.7 [33 to 85] | 63.8 [27 to 86] | 60.0 [28 to 80] | 59.3 [26 to 82] | 62.4 [26 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 8 | 7 | 13 | 38
  Male | 19 | 16 | 16 | 18 | 12 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 22 | 23 | 24 | 25 | 25 | 119
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Did Not Require Rescue Administration of Propofol to Achieve and Maintain Observer's Assessment of Alertness/Sedation (OAA/S) Score ≤4 During the Study Drug Administration.
Time Frame: Pre-dose, every 5 ± 2 minutes after start of study drug infusion and every 15 ± 2 minutes until 1 hour after study drug infusion. Before additional administration of sedative.
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Percentage of participants | 22.7 [7.8 to 45.4] | 13.0 [2.8 to 33.6] | 45.8 [25.6 to 67.2] | 68.0 [46.5 to 85.1] | 80.0 [59.3 to 93.2]
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; The closed testing procedure is used taking multiplicity into consideration, in which Dexmedetomidine 1.0 mcg/kg group, 0.5 mcg/kg group, 0.25 mcg/kg group, 0.067 mcg/kg group and the placebo group are tested in this order; Test type: Superiority; p < 0.001, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine 0.5 mcg/kg; Test type: Superiority; p = 0.003, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 3: Comparison: Placebo vs Dexmedetomidine 0.25 mcg/kg; Test type: Superiority; p = 0.086, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 4: Comparison: Placebo vs Dexmedetomidine 0.067 mcg/kg vs Dexmedetomidine 0.25 mcg/kg vs Dexmedetomidine 0.5 mcg/kg vs Dexmedetomidine 1.0 mcg/kg; Dose-response relationship is assessed using Mantel-extension test. In this analysis, dose of placebo group is hypothesized as 0 microg/kg. Dose-response relationship among Dexmedetomidine 4 dose groups excluding placebo group is also assessed using Mantel-extension test; Test type: Superiority; p < 0.001, Mantel-extension test; Stratified by the anesthesia type

2. Secondary Outcome: Number of Propofol Dosing Required to Achieve and Maintain OAA/S Score ≤4 During the Study Drug Administration
Time Frame: 15 minutes after the start of study drug, if the OAA/S score is 5.
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Number of dosing
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Number of dosing | 5.1 (4.7) | 3.7 (3.4) | 1.9 (2.3) | 0.8 (1.5) | 0.5 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine 0.5 mcg/kg; Test type: Superiority; p < 0.001, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 3: Comparison: Placebo vs Dexmedetomidine 0.25 mcg/kg; Test type: Superiority; p = 0.006, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 4: Comparison: Placebo vs Dexmedetomidine 0.067 mcg/kg; Test type: Superiority; p = 0.329, Mantel Haenszel; Stratified by the anesthesia type

3. Secondary Outcome: Dosage of Propofol Dosing Required to Achieve and Maintain OAA/S Score ≤4 During the Study Drug Administration
Time Frame: 15 minutes after the start of study drug, if the OAA/S score is 5.
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
mg/kg | 1.019 (0.933) | 0.744 (0.675) | 0.373 (0.459) | 0.166 (0.298) | 0.096 (0.231)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine 0.5 mcg/kg; Test type: Superiority; p < 0.001, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 3: Comparison: Placebo vs Dexmedetomidine 0.25 mcg/kg; Test type: Superiority; p = 0.006, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 4: Comparison: Placebo vs Dexmedetomidine 0.067 mcg/kg; Test type: Superiority; p = 0.371, Mantel Haenszel; Stratified by the anesthesia type

4. Secondary Outcome: Time to First Rescue Administration of Propofol
Time Frame: During the study drug infusion period (≥15 minutes [Approximate])
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
minutes | 25.5 [20.0 to 46.0] | 20 [20.0 to 22.0] | 24 [21.0 to NA] — The estimate dose not reach the point of 50%. | NA [61.0 to NA] — The estimate dose not reach the point of 50%. | NA [NA to NA] — The estimate dose not reach the point of 50%.
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log Rank; Stratified by the anesthesia type
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine 0.5 mcg/kg; Test type: Superiority; p = 0.001, Log Rank; Stratified by the anesthesia type
Statistical Analysis 3: Comparison: Placebo vs Dexmedetomidine 0.25 mcg/kg; Test type: Superiority; p = 0.212, Log Rank; Stratified by the anesthesia type

5. Secondary Outcome: Percentage of Patients Who Did Not Require Rescue Administration of Fentanyl During the Study Drug Administration
Time Frame: After the surgery start, the administration of fentanyl is permissible as required to treat pain. In case of repeated dose, the dosing interval should be ≥15 minutes.
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Percentage of participants | 95.5 [77.2 to 99.9] | 91.3 [72.0 to 98.9] | 100.0 [85.8 to 100.0] | 96.0 [79.6 to 99.9] | 96.0 [79.6 to 99.9]
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.869, Mantel Haenszel; Stratified by the anesthesia type

6. Secondary Outcome: Number of Fentanyl Dosing Required During the Study Drug Administration.
Time Frame: During the study drug administration
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Number of dosing
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Number of dosing | 0.1 (0.6) | 0.2 (0.7) | 0.0 (0.0) | 0.0 (0.2) | 0.1 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.897, Mantel Haenszel; Stratified by the anesthesia type

7. Secondary Outcome: Dosage of Fentanyl Dosing Required During the Study Drug Administration.
Time Frame: During the study drug administration
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
mcg/kg | 0.068 (0.320) | 0.085 (0.317) | 0.000 (0.000) | 0.018 (0.088) | 0.061 (0.304)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.897, Mantel Haenszel; Stratified by the anesthesia type

8. Secondary Outcome: Percentage of Time Spent OAA/S Score ≤4 During the Study Drug Infusion
Time Frame: as for outcome 1
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Percentage of time | 50.17 (23.88) | 58.15 (20.71) | 61.44 (18.28) | 70.07 (21.08) | 76.78 (14.07)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine 0.5 mcg/kg; Test type: Superiority; p = 0.002, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 3: Comparison: Placebo vs Dexmedetomidine 0.25 mcg/kg; Test type: Superiority; p = 0.116, Mantel Haenszel; Stratified by the anesthesia type

9. Secondary Outcome: Percentage of Time Spent OAA/S Score 3 to 4 During the Study Drug Infusion
Time Frame: as for outcome 1
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Percentage of time | 47.88 (25.31) | 56 (19.87) | 53.66 (17.5) | 65.3 (20.63) | 62.25 (23.14)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.088, Mantel Haenszel; Stratified by the anesthesia type

10. Secondary Outcome: Time to Attain the Point Where Patient is Recovered Assessed by Aldrete Score Following Discontinuation of the Study Drug Infusion
Time Frame: Every 15 ± 2 minutes until the score of each item becomes ≥1 and the total value becomes ≥8.
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Minutes | 15 [NA to NA] — There were a lot of tied values of the median in individual data, the 95% CI could not be calculated (could not become an interval). | 15 [NA to NA] — There were a lot of tied values of the median in individual data, the 95% CI could not be calculated (could not become an interval). | 15 [15.0 to 16.0] | 15 [NA to NA] — There were a lot of tied values of the median in individual data, the 95% CI could not be calculated (could not become an interval). | 15 [NA to NA] — There were a lot of tied values of the median in individual data, the 95% CI could not be calculated (could not become an interval).
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.085, Log Rank; Stratified by the anesthesia type

11. Secondary Outcome: Visual Analogue Scale (VAS) Score Evaluation by Investigator or Sub-investigator (Easiness of Maintenance of Sedation Level)
Description: VAS score ranges from 0 to 10, with 0 being the better/preferred outcome. Low values indicated more ease of maintenance of sedation level.
Time Frame: Within 24 hours after completion of the study drug administration
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 5.85 (3.54) | 4.36 (3.41) | 3.73 (3.19) | 2.81 (2.64) | 2.65 (2.98)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine 0.5 mcg/kg; Test type: Superiority; p = 0.014, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 3: Comparison: Placebo vs Dexmedetomidine 0.25 mcg/kg; Test type: Superiority; p = 0.055, Mantel Haenszel; Stratified by the anesthesia type

12. Secondary Outcome: Visual Analogue Scale (VAS) Score Evaluation by Investigator or Sub-investigator (Stability of Hemodynamic State)
Description: as for outcome 11
Time Frame: Within 24 hours after completion of the study drug administration
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 2.05 (2.21) | 3.3 (3.19) | 1.68 (1.46) | 1.72 (2.14) | 1.47 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.737, Mantel Haenszel; Stratified by the anesthesia type

13. Secondary Outcome: Visual Analogue Scale (VAS) Score Evaluation by Investigator or Sub-investigator (Stability of Respiratory State)
Description: as for outcome 11
Time Frame: Within 24 hours after completion of the study drug administration
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 2.35 (2.77) | 2.62 (2.79) | 1.8 (2.02) | 2.85 (2.9) | 3.12 (2.13)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.11, Mantel Haenszel; Stratified by the anesthesia type

14. Secondary Outcome: Visual Analogue Scale (VAS) Score Evaluation by Investigator or Sub-investigator (Subject's Cooperation)
Description: as for outcome 11
Time Frame: Within 24 hours after completion of the study drug administration
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 1.48 (1.67) | 1.8 (2.35) | 1.05 (1.46) | 1.15 (1.19) | 1.17 (1.46)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.567, Mantel Haenszel; Stratified by the anesthesia type

15. Secondary Outcome: Score Evaluation of Satisfaction and Anxiety of the Subject ("I Was Satisfied With This Anesthesia Procedure")
Description: Rating: 1 is the better/preferred value for scores from 1 to 4. Low values indicated more ease of maintenance of sedation level.
Time Frame: Within 24 hours after completion of the study drug administration (as much as possible)
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 1.7 (0.8) | 1.7 (1) | 1.2 (0.4) | 1.4 (0.7) | 1.3 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.044, Mantel Haenszel; Stratified by the anesthesia type
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine 0.5 mcg/kg; Test type: Superiority; p = 0.234, Mantel Haenszel; Stratified by the anesthesia type

16. Secondary Outcome: Score Evaluation of Satisfaction and Anxiety of the Subject ("I Did Not Feel Pain During the Surgery")
Description: as for outcome 15
Time Frame: Within 24 hours after completion of the study drug administration (as much as possible)
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 1.2 (0.7) | 1.2 (0.7) | 1.2 (0.7) | 1.4 (0.9) | 1.2 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.729, Mantel Haenszel; Stratified by the anesthesia type

17. Secondary Outcome: Score Evaluation of Satisfaction and Anxiety of the Subject ("If You May Undergo a Similar Surgery, the Same Anesthesia Procedure Will be Requested for the Next Time")
Description: as for outcome 15
Time Frame: Within 24 hours after completion of the study drug administration (as much as possible)
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 1.7 (1.1) | 1.5 (0.8) | 1.3 (0.6) | 1.5 (0.8) | 1.2 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.082, Mantel Haenszel; Stratified by the anesthesia type

18. Secondary Outcome: Score Evaluation of Satisfaction and Anxiety of the Subject ("Assess the Anxiety Level Before Surgery")
Description: Rating: 1 is the better/preferred value for scores from 1 to 5. Low values indicated more ease of maintenance of sedation level.
Time Frame: Within 24 hours after completion of the study drug administration (as much as possible)
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 2.2 (1.3) | 2.2 (1.3) | 2.2 (1.2) | 1.8 (1) | 2 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.451, Mantel Haenszel; Stratified by the anesthesia type

19. Secondary Outcome: Score Evaluation of Satisfaction and Anxiety of the Subject ("Assess the Anxiety Level During Surgery")
Description: as for outcome 18
Time Frame: Within 24 hours after completion of the study drug administration (as much as possible)
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 1.6 (1.1) | 1.6 (0.8) | 1.6 (0.9) | 1.4 (0.9) | 1.7 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.873, Mantel Haenszel; Stratified by the anesthesia type

20. Secondary Outcome: Score Evaluation of Satisfaction and Anxiety of the Subject ("Assess the Anxiety Level After Surgery")
Description: as for outcome 18
Time Frame: Within 24 hours after completion of the study drug administration (as much as possible)
Population: Full Analysis Set<FAS>: FAS is defined as all patients who were administered with the study drugs.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
Number analyzed (Participants) | 22 | 23 | 24 | 25 | 25
Scores on a scale | 1.6 (0.9) | 1.6 (1) | 1.6 (0.6) | 1.3 (0.7) | 1.5 (1)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine 1.0 mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.374, Mantel Haenszel; Stratified by the anesthesia type

ADVERSE EVENTS:
Time Frame: Adverse events that occurred from the start of treatment to 24 hours after the end of treatment, a median of 67 - 87 mins treatment depending on treatment arms.
Arm/Group | Placebo | Dexmedetomidine 0.067 mcg/kg | Dexmedetomidine 0.25 mcg/kg | Dexmedetomidine 0.5 mcg/kg | Dexmedetomidine 1.0 mcg/kg
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/24 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/23 | 0/24 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 19/22 | 21/23 | 24/24 | 22/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Dexmedetomidine 0.067 mcg/kg (N=23) | Dexmedetomidine 0.25 mcg/kg (N=24) | Dexmedetomidine 0.5 mcg/kg (N=25) | Dexmedetomidine 1.0 mcg/kg (N=25)
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Dexmedetomidine 0.067 mcg/kg (N=23) | Dexmedetomidine 0.25 mcg/kg (N=24) | Dexmedetomidine 0.5 mcg/kg (N=25) | Dexmedetomidine 1.0 mcg/kg (N=25)
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headaches (Nervous system disorders) | 2 | 1 | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 8 | 11 | 9 | 10 | 11
Tachycardia (Cardiac disorders) | 2 | 3 | 0 | 0 | 0
Vasculitides (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 5 | 2 | 2 | 3 | 8
Hypotension (Vascular disorders) | 5 | 12 | 11 | 8 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 12 | 10 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 3 | 3
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Glossoptosis (Gastrointestinal disorders) | 3 | 0 | 0 | 2 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Erythemas (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0
Bladder irritation (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 1 | 0 | 0
Puncture site pain (General disorders) | 2 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator publishes any results of this study, a pre-publication manuscript shall be provided the sponsor for review at least 60 days prior to the submission of the manuscript to the publisher.